CLINICAL TRIAL: NCT04275297
Title: Optimizing Psychosocial Treatment of Interstitial Cystitis/Bladder Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lindsey Mckernan, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 193461; K23DK118118 (NIH)
Record Dates: First submitted 2020-02-11; First posted 2020-02-19 (Actual); Results first posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Chronic Interstitial Cystitis; Bladder Pain Syndrome; Cystitis, Interstitial; Painful Bladder Syndrome; Cystitis, Chronic Interstitial; Interstitial Cystitis; Interstitial Cystitis, Chronic; Interstitial Cystitis (Chronic) With Hematuria; Interstitial Cystitis (Chronic) Without Hematuria; Chronic Prostatitis; Chronic Prostatitis With Chronic Pelvic Pain Syndrome
Keywords: interstitial cystitis; bladder pain syndrome; clinical trial; psychosocial intervention; pelvic pain; therapy; urological chronic pelvic pain syndrome; chronic prostatitis; self-management; cognitive behavioral therapy
MeSH Terms: conditions — Cystitis, Interstitial; Bronchiolitis Obliterans Syndrome; Prostatitis; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: The study involves a two group parallel design, with one group receiving individual psychosocial intervention online/in person and another individual symptom monitoring and discussion via telephone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial Treatment (Experimental): The psychosocial self-management intervention consists of 8 weekly 50-minute individual visits with an assigned trained therapist. Sessions follow a structured protocol that has been developed with the patient population. Treatment modules are individualized and include topics such as pain coping strategies, relaxation training, education on IC/BPS, and communication strategies.
  Interventions: Behavioral: Psychosocial Treatment
- Attention Control (Placebo Comparator): The attention control condition consists of 8 weekly telephone calls with a study interventionist. Sessions will occur via scheduled telephone calls and follow a structured procedure. Telephone calls are designed to monitor symptoms and overall wellness. Each week, participants will be asked about current symptoms, flare patterns, and physical and emotional wellbeing.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Psychosocial Treatment — The psychosocial intervention will consist of 8 weekly 50-minute individual visits with the assigned therapist.
  Arms: Psychosocial Treatment
Behavioral: Attention Control — The Attention Control will reflect a similar visit pattern and duration as intervention sessions.
  Arms: Attention Control

SUMMARY:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a severe pain condition affecting 3-8 million people in the United States lacking treatments that work. Emotional suffering is common in IC/BPS and known to make physical symptoms worse, and studies show patient sub-groups respond differently to treatment. By creating and testing a psychosocial intervention specific to IC/BPS, we will learn if this intervention improves patient wellness, who the intervention works best for, and how the body's pain processing influences outcomes.

DETAILED DESCRIPTION:
Interstitial cystitis/bladder pain syndrome (IC/BPS) is a debilitating, incurable, and costly pain condition affecting approximately 3-8 million individuals in the United States and is extremely challenging to treat. Evidence suggests psychosocial factors accompany and intensify the illness.

Unaddressed psychosocial co-morbidities are associated with reduced functionality and poorer outcomes, which suggests that psychosocial symptoms and bladder-specific symptoms reinforce each other. While psychosocial self-management interventions have demonstrated efficacy for other pain conditions, the IC/BPS field lacks the gold standard - randomized controlled trials - studying these interventions. At the same time, the chronic pain field is adopting a new approach driven by mechanisms of illness and treatment. Growing evidence suggests that subgroups (called "phenotypes") of patients with IC/BPS respond differently to medical intervention. Presence of central sensitization (CS) largely defines patient subgroups and may be a biological factor affecting response to medical treatment. The overall goal of this project is to fully develop, optimize, and evaluate a patient-centered CBT self-management intervention specific to IC/BPS. To achieve this goal, we will develop (Aim 1) and test (Aim 2) an empirically-based psychosocial treatment for IC/BPS compared to attention control, while examining pain mechanisms and subgroup characteristics that may alter treatment response (Aim 3). We hypothesize that a) inclusion of a self-management intervention will be more effective than a control treatment for IC/BPS, and that b) treatment effects will be moderated by degree of psychological co-morbidity, presence of chronic overlapping pain conditions, and elevated central sensitization. Successful completion of these aims will determine whether the addition of a tailored self-management intervention for IC/BPS will improve outcomes compared to control, whether particular subgroups are more responsive to this intervention, and whether a biological mechanism (CS) influences treatment responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of IC/BPS as given by providers or indicated by assessments

Exclusion Criteria:

* Comorbid neurological conditions including spinal cord injury or systematic neurologic illnesses, or central nervous system diseases such as brain tumor or stroke
* Current or history of diagnosis of primary psychotic or major thought disorder within the past five years
* Hospitalization for psychiatric reasons other than suicidal ideation, homicidal ideation, and/or PTSD (within the past 5 years)
* Psychiatric or behavioral conditions in which symptoms are unstable or severe (e.g. current delirium, mania, psychosis, suicidal ideation, homicidal ideation, substance abuse dependency) reported within the past six months
* Non-English speaking
* Presenting symptoms at time of screening that would interfere with participation, specifically active suicidal ideation with intent to harm oneself or active delusional or psychotic thinking
* Difficulties or limitations communicating over the telephone
* Any planned life events that would interfere with participating in the key elements of the study
* Any major active medical issues that could preclude participation
* Currently being treated for cancer
* Cancer-related pain
* Currently engaged in individual counseling/psychotherapy or unwilling to pause this treatment for the trial duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey McKernan, PhD MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This study is occurring via a career development award mechanism through the NIDDK. The PI will establish an IPD sharing plan following consultation with study team mentors at a bi-annual mentorship team meeting in April. The information will be updated in the system accordingly.

REFERENCES:
- [Background] Hanno PM, Burks DA, Clemens JQ, Dmochowski RR, Erickson D, Fitzgerald MP, Forrest JB, Gordon B, Gray M, Mayer RD, Newman D, Nyberg L Jr, Payne CK, Wesselmann U, Faraday MM; Interstitial Cystitis Guidelines Panel of the American Urological Association Education and Research, Inc. AUA guideline for the diagnosis and treatment of interstitial cystitis/bladder pain syndrome. J Urol. 2011 Jun;185(6):2162-70. doi: 10.1016/j.juro.2011.03.064. Epub 2011 Apr 16. PMID 21497847
- [Background] Berry SH, Bogart LM, Pham C, Liu K, Nyberg L, Stoto M, Suttorp M, Clemens JQ. Development, validation and testing of an epidemiological case definition of interstitial cystitis/painful bladder syndrome. J Urol. 2010 May;183(5):1848-52. doi: 10.1016/j.juro.2009.12.103. Epub 2010 Mar 29. PMID 20303099
- [Background] Brummett CM, Bakshi RR, Goesling J, Leung D, Moser SE, Zollars JW, Williams DA, Clauw DJ, Hassett AL. Preliminary validation of the Michigan Body Map. Pain. 2016 Jun;157(6):1205-1212. doi: 10.1097/j.pain.0000000000000506. PMID 26835782
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB. Fibromyalgia criteria and severity scales for clinical and epidemiological studies: a modification of the ACR Preliminary Diagnostic Criteria for Fibromyalgia. J Rheumatol. 2011 Jun;38(6):1113-22. doi: 10.3899/jrheum.100594. Epub 2011 Feb 1. PMID 21285161
- [Background] Kratz AL, Schilling SG, Goesling J, Williams DA. Development and initial validation of a brief self-report measure of cognitive dysfunction in fibromyalgia. J Pain. 2015 Jun;16(6):527-36. doi: 10.1016/j.jpain.2015.02.008. Epub 2015 Mar 4. PMID 25746197
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Desrochers G, Bergeron S, Khalife S, Dupuis MJ, Jodoin M. Fear avoidance and self-efficacy in relation to pain and sexual impairment in women with provoked vestibulodynia. Clin J Pain. 2009 Jul-Aug;25(6):520-7. doi: 10.1097/AJP.0b013e31819976e3. PMID 19542801
- [Background] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Background] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Rampakakis E, Ste-Marie PA, Sampalis JS, Karellis A, Shir Y, Fitzcharles MA. Real-life assessment of the validity of patient global impression of change in fibromyalgia. RMD Open. 2015 Sep 14;1(1):e000146. doi: 10.1136/rmdopen-2015-000146. eCollection 2015. PMID 26535150
- [Background] Sherman AL, Morris MC, Bruehl S, Westbrook TD, Walker LS. Heightened Temporal Summation of Pain in Patients with Functional Gastrointestinal Disorders and History of Trauma. Ann Behav Med. 2015 Dec;49(6):785-92. doi: 10.1007/s12160-015-9712-5. PMID 25967582
- [Background] Starkweather AR, Heineman A, Storey S, Rubia G, Lyon DE, Greenspan J, Dorsey SG. Methods to measure peripheral and central sensitization using quantitative sensory testing: A focus on individuals with low back pain. Appl Nurs Res. 2016 Feb;29:237-41. doi: 10.1016/j.apnr.2015.03.013. Epub 2015 Apr 8. PMID 26856520
- [Background] Li J, Simone DA, Larson AA. Windup leads to characteristics of central sensitization. Pain. 1999 Jan;79(1):75-82. doi: 10.1016/S0304-3959(98)00154-7. PMID 9928779
- [Background] Shy ME, Frohman EM, So YT, Arezzo JC, Cornblath DR, Giuliani MJ, Kincaid JC, Ochoa JL, Parry GJ, Weimer LH; Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Quantitative sensory testing: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2003 Mar 25;60(6):898-904. doi: 10.1212/01.wnl.0000058546.16985.11. PMID 12654951
- [Background] Ezenwa MO, Molokie RE, Wang ZJ, Yao Y, Suarez ML, Pullum C, Schlaeger JM, Fillingim RB, Wilkie DJ. Safety and Utility of Quantitative Sensory Testing among Adults with Sickle Cell Disease: Indicators of Neuropathic Pain? Pain Pract. 2016 Mar;16(3):282-93. doi: 10.1111/papr.12279. Epub 2015 Jan 12. PMID 25581383

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psychosocial Treatment | Attention Control
Started | 52 | 26
Completed Optional In-person Assessment Including Quantitative Sensory Testing | 29 | 11
Completed | 51 | 25
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: One participant enrolled in the study and was randomized to attention control, but did not complete any baseline assessments. This participant's age was accessible from the consent form, and was therefore included in that baseline measurement, but no other data from this participant was gathered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychosocial Treatment | Attention Control | Total
Number analyzed (Participants) | 52 | 26 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (16.5) | 43.1 (16) | 44.4 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant was enrolled in the study and randomized to attention control, but did not complete any baseline assessments. This participant's age was accessible from the consent form so was included in that baseline measurement, but no other baseline data was gathered from this participant.
  Participants
    number analyzed (Participants) | 52 | 25 | 77
    Female | 48 | 23 | 71
    Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant was enrolled in the study and randomized to attention control, but did not complete any baseline assessments. This participant's age was accessible from the consent form so was included in that baseline measurement, but no other baseline data was gathered from this participant.
  Participants
    number analyzed (Participants) | 52 | 25 | 77
    Hispanic or Latino | 1 | 0 | 1
    Not Hispanic or Latino | 51 | 25 | 76
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One participant was enrolled in the study and randomized to attention control, but did not complete any baseline assessments. This participant's age was accessible from the consent form so was included in that baseline measurement, but no other baseline data was gathered from this participant.
  Participants
    number analyzed (Participants) | 52 | 25 | 77
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 2 | 1 | 3
    White | 49 | 21 | 70
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 52 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change in the Genitourinary Pain Index (GUPI) 2 Months
Description: The Genitourinary Pain Index measures genitourinary symptom severity in both men and women. It is comprised of three subscales: pain, urinary symptoms, and impact on quality of life. The total score ranges from 0-35, with 0 being the lowest severity of symptoms and 35 being the highest.
Time Frame: baseline to 2 months
Population: We analyzed a total of N=77 individuals from baseline to post-treatment. Below is the change in the total genitourinary pain index (GUPI) score between both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 52 | 25
score on a scale | 6.6 (6.9) | 4.8 (9.0)

2. Primary Outcome: Change in the Genitourinary Pain Index (GUPI) 5 Months
Description: as for outcome 1
Time Frame: baseline to 5 months
Population: We analyzed a total of N=77 individuals from baseline to follow-up. Below is the change in the total genitourinary pain index (GUPI) score between both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 52 | 25
score on a scale | 8.1 (9.9) | 6.6 (7.3)

3. Secondary Outcome: Change in Depressive Symptoms Measured by the Patient Health Questionnaire (PHQ-8)
Description: The eight-item Patient Health Questionnaire depression scale (PHQ-8) is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies. It consists of 8 questions where participants indicate on a Likert scale the extent to which they have experienced symptoms of depression within the past two weeks, with 0 being "not at all" and 3 being "nearly every day." Cumulative scores range from 0-24, with cutoff points for none, mild, moderate, moderately severe, and severe marked at 5, 10, 15, and 20.
Time Frame: baseline, 2 months (after treatment is complete), 5 months
Population: We analyzed a total of N=77 individuals from baseline to post-treatment. Below is the change in the total PHQ score between both timepoints both from pre-post treatment and then from pre-treatment to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 52 | 25
score on a scale
  Baseline to post-treatment (2 months) | 0.9 (4.6) | 1.0 (4.3)
  Baseline to follow-up (5 months) | 0.8 (5.2) | 0.0 (3.4)

4. Secondary Outcome: The Widespread Pain Index (Derived From CHOIR Bodymap)
Description: The Widespread Pain Index measures the location(s) of chronic pain complaints and widespread body pain. Widespread pain was assessed using the Collaborative Health Outcomes Information Registry (CHOIR) bodymap, condensed into a Widespread Pain Index (WPI) score assessing 19 potential body pain areas. Scores on the WPI range from 0-19, with one point given for each potential body pain area endorsed; higher scores indicate higher widespread pain. The WPI was coupled with the Fibromyalgia Symptom Scale (FSS) below, a 7-item questionnaire, to calculate the American College of Rheumatology classification criteria for fibromyalgia, and assess fibromyalgia symptom severity (higher scores indicate higher symptom severity). The WPI total (0-19) can be combined with the FSS (0-12) in a sum total score (0-31) to assess the degree of a person's widespread pain and fibromyalgia symptom severity, with higher scores indicating a worse outcome.
Time Frame: baseline, 2 months (after treatment is complete), 5 months
Population: We analyzed a total of N=77 individuals from baseline to follow-up. Below is the change in the total WPI score between both timepoints both from pre-post treatment and then from pre-treatment to follow-up. Change in total FSS score is not included here, but is reported separately.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 52 | 25
score on a scale
  Baseline to post treatment (2 months) | 0.6 (2.9) | 0.1 (2.7)
  Baseline to follow up (5 months) | 0.9 (3.5) | 0.4 (3.6)

5. Secondary Outcome: Fibromyalgia Symptom Scale (FSS)
Description: 7-item questionnaire assessing modified 2010 American College of Rheumatology diagnostic criteria for fibromyalgia and includes a) an index of widespread pain and b) an index of symptom severity via patient self-report. The FSS is the index of symptom severity and can range from 0-12. Higher scores indicate higher symptom severity, a worse outcome. When combined with the WPI score above, a total score on this scale (WPI + FSS) ranges from 0-31, with scores ≥ 13 indicating a high likelihood of fibromyalgia.
Time Frame: baseline, 2 months (after treatment is complete), 5 months
Population: We analyzed a total of N=77 individuals from baseline to post-treatment. Below is the change in the total FSS score between both timepoints both from pre-post treatment and then from pre-treatment to follow-up. Change in WPI is reported separately above.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 52 | 25
score on a scale
  Baseline to post treatment (2 months) | 0.4 (1.9) | 0.7 (1.4)
  Baseline to follow-up (5 months) | 0.8 (1.8) | 0.2 (1.3)

6. Secondary Outcome: Change in Posttraumatic Stress Symptoms Measured by PTSD Checklist for DSM-5 (PCL-5) With Criterion A
Description: The PTSD Checklist for the DSM-5 measures post-traumatic stress. It utilizes the symptom checklist for PTSD in the DSM-5 and inquires about trauma-induced thoughts and behaviors in the past month. The total score ranges from 0-80, with 31-33 and above indicating probable diagnosis of PTSD.
Time Frame: baseline, 2 months (after treatment is complete), 5 months
Population: We analyzed a total of N=77 individuals from baseline to post-treatment. Below is the change in the total PCL-5 score between both timepoints both from pre-post treatment and then from pre-treatment to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 52 | 25
score on a scale
  Baseline to post-treatment (2 months) | -2.8 (9.9) | -1.3 (11.6)
  Baseline to follow-up (5 months) | 0.1 (13.8) | -3.5 (12.1)

7. Secondary Outcome: Change in Anxiety Symptoms Measured by the Generalized Anxiety Disorder (GAD-7) Questionnaire
Description: The Generalized Anxiety Disorder (GAD-7) questionnaire is a self-administered 7 item instrument that uses some of the DSM-V criteria for GAD to identify probable cases of GAD along with measuring anxiety symptom severity. Questions are on a 4-point Likert scale, with 0 being "not at all sure" and 3 being "nearly every day." Cumulative scoring is tiered from minimal anxiety (0-4) to mild anxiety (5 to 9) to moderate anxiety (10-14) to severe anxiety (15-21).
Time Frame: baseline, 2 months (after treatment is complete), 5 months
Population: We analyzed a total of N=77 individuals from baseline to post-treatment. Below is the change in the total GAD-7 score between both timepoints both from pre-post treatment and then from pre-treatment to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 52 | 25
score on a scale
  Baseline to post-treatment (2 months) | 0.5 (4) | 0.6 (4)
  Baseline to follow-up (5 months) | 0.1 (4.5) | -0.1 (3.5)

8. Secondary Outcome: Difference in Response to Treatment/Perceived Improvement and Quality of Life Between Groups as Measured by the Patient Global Impression of Change Scale (PGIC)
Description: Patient Global Impression of Improvement measures the response of a condition to an intervention. Patients rate their impression of change on a Likert scale ranging from 1-7 with 1 being "No change/condition has gotten worse" to 7 being "a great deal better and a considerable improvement that has made all the difference." This scale was administered at post-treatment and follow-up only.
Time Frame: 2 months (after treatment is complete), 5 months
Population: We analyzed a total of N=77 individuals from baseline to post-treatment. Below is the change in the total PGIC score between both timepoints both from pre-post treatment and then from pre-treatment to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 52 | 25
score on a scale
  Baseline to post-treatment (2 months) | 4.7 (1.6) | 2.8 (1.6)
  Baseline to follow-up (5 months) | 4.4 (1.5) | 3.1 (1.6)

9. Secondary Outcome: Quantitative Sensory Testing (Optional) - Threshold Average
Description: Psychophysical testing methods replicated existing protocols used at VUMC and include the following elements: 1) an evaluation of temporal summation (as a biomarker for central sensitization), 2) thermal pain threshold and tolerance. Thermal measures involved four pain threshold trials, followed by four pain tolerance trials, with the probe applied to slightly different target sites for each trial to avoid local sensitization. Means for the four threshold and tolerance trials are separately derived, and threshold is reported here. Scores range from 0 = "No Pain or Warmth" to 100 = "Worst Possible Pain", with higher scores indicating a higher pain threshold.
Time Frame: baseline
Population: We analyzed a total of 40 participants who completed Quantitative Sensory Testing at baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 29 | 11
score on a scale | 44.65 (3.41) | 40.76 (2.96)

10. Secondary Outcome: Quantitative Sensory Testing (Optional) - Tolerance Average
Description: Psychophysical testing methods replicated existing protocols used at VUMC and include the following elements: 1) an evaluation of temporal summation (as a biomarker for central sensitization), 2) thermal pain threshold and tolerance. Thermal measures involved four pain threshold trials, followed by four pain tolerance trials, with the probe applied to slightly different target sites for each trial to avoid local sensitization. Means for the four threshold and tolerance trials are separately derived, and tolerance is reported here. Scores range from 0 = "No Pain or Warmth" to 100 = "Worst Possible Pain", with higher scores indicating a higher pain tolerance.
Time Frame: baseline
Population: We analyzed a total of 40 participants who completed Quantitative Sensory Testing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 29 | 11
units on a scale | 47.89 (1.09) | 47.29 (1.79)

11. Secondary Outcome: Quantitative Sensory Testing - Temporal Summation (Slope)
Description: Psychophysical testing methods will replicate existing protocols used at VUMC and include the following elements: 1) an evaluation of temporal summation (as a biomarker for central sensitization), 2) thermal pain threshold and tolerance. Regarding temporal summation: in each sequence, immediately after each heat pulse, subjects provide a verbal numeric pain intensity rating on a 0-100 scale (0 = "No Pain or Warmth" and 100 = "Worst Possible Pain"). The standardized slope of the line fitted to the series of 10 pulses at each temperature indexes temporal summation and serves as a quantitative marker of central sensitization. These slopes reflected the relationship between pain and pulse, representing average pain increase for each unit increase in pulse.
Time Frame: Baseline
Population: A total of 40 participants completed (optional) quantitative sensory testing at baseline allowing us to calculate temporal summation.
Measure: Mean (Standard Deviation); unit: units on a scale/pulse
Arm/Group | Psychosocial Treatment | Attention Control
Number analyzed (Participants) | 29 | 11
units on a scale/pulse | -.23 (2.18) | -.21 (2.70)

ADVERSE EVENTS:
Time Frame: From date of randomization up to 97 days post-treatment, an average of 5.5 months.
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. Adverse events were collected from the time of randomization through participant completion.
Arm/Group | Psychosocial Treatment | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/26
Other Adverse Events (participants affected / at risk) | 1/52 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychosocial Treatment (N=52) | Attention Control (N=26)
Temporary pain increase (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Participant experienced exacerbation of pre-existing pelvic pain following administration of quantitative sensory testing protocol. Participant reported pain exacerbation for approximately two hours.

LIMITATIONS AND CAVEATS:
As this trial was conducted at the outset of the COVID-19 pandemic, the psychological intervention that was planned for in-person sessions transitioned entirely to telehealth for the duration of the study. Second, the in-person assessment which included quantitative sensory testing was made optional.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT04275297/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT04275297/ICF_001.pdf